CLINICAL TRIAL: NCT03862378
Title: Prediction of Intra-abdominal Infectious Complication by Drainage Fluid Analysis After Gastrointestinal Cancer Surgery
Brief Title: Prediction of Intra-abdominal Infectious Complication by Drainage Fluid Analysis
Acronym: APPEAL-GC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Ziyu Li, MD, Professor, Peking University
Other Study IDs: 2016YJZ32
Record Dates: First submitted 2019-01-31; First posted 2019-03-05 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Complication; Anastomotic Leak; Intraabdominal Infections; Inflammatory Response; Gastrointestinal Cancer
MeSH Terms: conditions — Anastomotic Leak; Intraabdominal Infections; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples Without DNA — In this study, we will collect the discarded drainage fluid for each patient for further analysis. The samples will be collected and stored in -80 refrigerators until analysis. The candidate targets include IL-1, IL-6, IL-10, TNF-a, MMP2, MMP9.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group One: All patients underwent gastric or colorectal cancer surgery in the participating centers will be included. Clinical data, drainage cytokine levels will be recorded.

SUMMARY:
In our previous study, a nomogram model was established to predict intra-abdominal infectious complications after gastrointestinal surgery. This model was based on the clinical data and the drainage fluid cytokine levels, and it received an AUC >0.9. In this study, validation of this nomogram is planned to be conducted in this prospective cohort study.

DETAILED DESCRIPTION:
Intra-abdominal infectious complications such as anastomotic leakage are the most feared but common complications after gastrointestinal surgery. In our previous study, a nomogram model was established to predict intra-abdominal complications after gastrointestinal surgery. This model was based on the clinical data and the drainage fluid cytokine levels, and it received an AUC >0.9. A predicting score (i.e. APPEAL-GC score) was created based on the model. In this study, validation of this score in predicting intra-abdominal complications is planned to be conducted in this prospective cohort study.

In this study, all patients undergoing gastric or colorectal cancer surgery with a primary anastomosis will be included. The clinical data and complication data will be prospectively collected; the discarded drainage fluid will be collected and analyzed afterward. No additional intervention will be applied.

The cytokine levels in the drainage fluid will be evaluated, and together with the clinical data, an APPEAL-GC score will be created for each patient. We will investigate whether the above-mentioned score is able to predict the intraabdominal complications after surgery. The predictive value (clinical usefulness) of the score will be validated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Planned surgery for gastric or colorectal cancer with primary anastomosis.
* Inform consent signed before surgery.

Exclusion Criteria:

* No drainage tube placed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational study intends to include all patients undergoing gastric or colorectal cancer with primary anastomosis. Because drainage fluid analysis is necessary for the prediction model, patients without the tube will be excluded.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive value of the nomogram prediction model (APPEAL-GC score) | From surgery until discharge, up to 90 days.
  The positive predictive value of the APPEAL-GC score in predicting the intra-abdominal infectious complications. Intra-Abdominal infectious complications include anastomotic leakage and other abdominal infectious complications. The complication definitions are in accordance with the Chinese consensus of gastrointestinal complication diagnosis and registration.
  The APPEAL-GC score was derived from our recently finished study (unpublished). It includes evaluation of the surgical type (open or laparoscopic), resection range, age, and cytokine levels on the postoperative day 3. A score of each patient can be determined, and a pre-set cut-off value (unpublished data) was determined in our previous study based on the AUC analysis.
  In this study, each patient will be scored accordingly. The positive predictive value and negative predictive value of the cut-off value will be evaluated.

SECONDARY OUTCOMES:
Abdominal infection rate. | From surgery until discharge, up to 90 days.
  Number of anastomotic leak and other abdominal infection patients divided by the total inclusions.
Abdominal infection outcome. | From surgery until discharge, up to 90 days.
  It is categorized as cured, not cured at discharge, death. The doctor is required to select one option at patient discharge. Proportions of different outcomes will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Ziyu Li, MD PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided